CLINICAL TRIAL: NCT00116233
Title: Peds. Multicenter Study
Brief Title: Pediatric Multicenter Study of REPEL-CV
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: SyntheMed (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LMS0104RCV
Record Dates: First submitted 2005-06-27; First posted 2005-06-28 (Estimated); Last update posted 2005-06-28 (Estimated); Status verified 2005-06

CONDITIONS: Adhesions
Keywords: post operative adhesions
MeSH Terms: conditions — Tissue Adhesions

INTERVENTIONS:
Device: REPEL-CV

SUMMARY:
This trial will study REPEL-CV for reducing post operative adhesions following cardiovascular (cv) surgery.

DETAILED DESCRIPTION:
- Efficacy at second sternotomy

ELIGIBILITY:
Inclusion Criteria:

* Stage sternotomies

Exclusion Criteria:

* Delayed closure beyond 5 days

Ages: 1 Day to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child

CONTACTS AND LOCATIONS:
Overall Officials: Eli Pines, Study Director — SyntheMed
Locations (1):
- SyntheMed, Little Silver, New Jersey, United States